CLINICAL TRIAL: NCT04006314
Title: Exploring the Effectiveness of Simultaneous Autologous Platelet Rich Plasma and Neural Prolotherapy Injections in Treating Patients With Moderate to Severe Degrees of Knee Osteoarthritis
Brief Title: Platelet Rich Plasma and Neural Prolotherapy Injections in Treating Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Carl P.C. Chen, Director, Department of Physical Medicine & Rehabilitation, Chang Gung Memorial Hospital
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201701924A3
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Knee Osteoarthritis
Keywords: platelet rich plasma; neural prolotherapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients are divided into two groups. One group receiving PRP injections only. One group receiving PRP plus neural prolotherapy injections.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving PRP injections or PRP plus neural prolotherapy (Other): PRP injection into the knee joint and pes anserinus complex. Dextrose solution to the genicular nerves.
  Interventions: Other: Autologous platelet rich plasma and dextrose solution.

INTERVENTIONS:
Other: Autologous platelet rich plasma and dextrose solution. — Autologous platelet rich plasma are injected into the knee joint and pes anserinus complex.
  Dextrose solutions are injected to the genicular nerves.

SUMMARY:
Osteoarthritis (OA) of the knees is the most common degenerative disorder seen in a rehabilitation outpatient clinic. It is characterized by metabolic, biochemical, and structural changes in the articular cartilage and the surrounding tissues. Knee OA patients are often troubled with knee pain and functional disturbance. Several studies have shown that the earlier the injection of autologous platelet rich plasma (a PRP) to treat early stages of knee OA, the better the treatment outcome. However, no consensus has been reached as to whether PRP injection is beneficial for patients with moderate to severe degrees of knee OA. Studies have also shown that the application of neural prolotherapy (NPT) to the genicular nerves may have beneficial effects in treating patients with severe knee OA. However, patients may start to walk for a longer period of time due to reduced knee pain after NPT. If the regenerative effect of PRP is not yet obvious on the knee cartilage, this excess walking may result in further destruction of the knee joints. No studies have examined the combined treatment effect of a PRP and NPT on patients with moderate to severe degrees of knee OA.

NPT is the injection of low percentage dextrose water (5%) with the rationale to repair and reduce pain caused by the nerves. We would like to bring our PRP study to a higher level by conducting a two-year study to recruit patients with moderate to severe degrees of knee OA. PRP will be injected into the knee joint and the pes anserine tendons. Simultaneous NPT will also be performed to the genicular nerves. The effectiveness will be examined using proteomics, isokinetic measurements and functional scale evaluations. Synovial fluid (SF) is in direct contact with the cartilage and synovium, protein biomarkers related to the disease pathophysiology of knee OA are contained within the SF and will be used for proteomic analysis. Patients will receive monthly injections for a total of 3 months. In short, if inflammatory proteins in the SF are not reduced after PRP injections, this indicates that PRP is not a good treatment choice for patients with moderate to severe degrees of knee OA. If inflammatory protein concentrations are further increased after NPT as patients may start strenuous exercises with reduced knee pain, more knee joint destruction may result.

DETAILED DESCRIPTION:
Patients will receive monthly injections for a total of 3 months. In short, if inflammatory proteins in the SF are not reduced after PRP injections, this indicates that PRP is not a good treatment choice for patients with moderate to severe degrees of knee OA. If inflammatory protein concentrations are further increased after NPT as patients may start strenuous exercises with reduced knee pain, more knee joint destruction may result. This signifies that NPT has pain reduction effect only and is not a viable treatment option. Roentgenograms may not show immediate signs of increased degeneration on the knee joints, but SF proteomic findings can provide us with evidences suggesting whether there is ongoing knee joint destruction. Upon the completion of this study, adequate scientific evidences will be gathered to know whether simultaneous PRP and NPT injections is a feasible option in treating patients with moderate to severe degrees of knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffered from chronic unilateral knee pain for more than 4 months and with roentgenogram degenerative findings of grades 3 and 4 on the Kellgren-Lawrence Classification of Osteoarthritis scale (meaning moderate to severe degrees of knee OA) will be recruited.
2. The volume of the SF in the supra-patellar bursa region is enough (at least 2 mm thickness in bursa fluid as measured by ultrasound) to be aspirated via ultrasound guidance.
3. Small volume of SF will be aspirated first and sent for SF analysis. SF showing evidences of crystals suggesting possible gouty arthritis and infection will not be included in this study.
4. Patient has previously received oral NSAIDs and physical modality treatments but WITHOUT any obvious improvements in knee pain and function.
5. The usage of musculoskeletal ultrasound to confirm that the supra-patellar bursa is in communication with the synovial cavity of the knee joint. This is to prevent the aspiration of isolated cystic lesion at the supra-patellar region.

Exclusion Criteria:

1. Total obliteration of knee joint as shown on the roentgenogram images.
2. Patient has systemic disorders such as diabetes, rheumatoid arthritis, major axial deviation of the knee joint (varus >5°, valgus >5°), hematological diseases (coagulopathy), severe cardiovascular diseases, infections, and immune-depression.
3. Patients in therapy with anticoagulants, and taking NSAIDs within the 5 days before blood harvest.
4. Patients with hemoglobin value of less than 11 g/dl, and platelet counts of less than 150,000/mm3.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Lequesne knee osteoarthritis questionnaire | About 10 minutes are required to evaluate the score of LeQuesne index.
  Lequesne knee osteoarthritis functional index which includes distance, pain, and function.
Two-dimensional electrophoresis (proteomics) | Two days are required to measure the protein band intensities on the gels.
  Hundreds of protein spots can be viewed on 2-dimensional electrophoresis gels. The intensity of each spot represents protein concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Carl P.C. Chen, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No